CLINICAL TRIAL: NCT03163121
Title: Safety and Protective Efficacy of Genetically Attenuated Pf∆b9∆Slarp (PfSPZ-GA1) Malaria Parasites in Healthy Dutch Volunteers
Brief Title: Safety and Protective Efficacy of Genetically Attenuated PfSPZ-GA1 Vaccine in Healthy Dutch Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Radboud University Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GA1; NL56657.000.16 (Other: ToetsingOnline); 2016-000893-39 (EudraCT Number)
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; PfSPZ Vaccine; PfSPZ-GA1 Vaccine; Controlled human malaria infection (CHMI); Genetically attenuated sporozoites; Plasmodium falciparum sporozoites (PfSPZ)
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage A is an open label study. Stage B of the clinical study will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group 1 - PfSPZ-GA1 Vaccine (Experimental): Group 1 will comprise of 3 volunteers who will receive one immunization of 1.35 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine via DVI.
  Volunteers will be followed closely for monitoring of adverse events and possible breakthrough blood infections by testing for the presence of parasitemia by qPCR. All volunteers will be treated with a curative regimen of atovaquone/proguanil (A/P) should break-through parasites be detected in the peripheral blood, or at the end of the follow-up period (28 days) if they are not qPCR positive. Six months after the inoculation, a final visit will take place to assess adverse events.
  Interventions: Biological: PfSPZ-GA1 Vaccine
- Group 2 - PfSPZ-GA1 Vaccine (Experimental): Group 2 will comprise of 3 volunteers who will receive one immunization of 4.5 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine via DVI.
  Volunteers will be followed closely for monitoring of adverse events and possible breakthrough blood infections by testing for the presence of parasitemia by qPCR. All volunteers will be treated with a curative regimen of atovaquone/proguanil (A/P) should break-through parasites be detected in the peripheral blood, or at the end of the follow-up period (28 days) if they are not qPCR positive. Six months after the inoculation, a final visit will take place to assess adverse events.
  Interventions: Biological: PfSPZ-GA1 Vaccine
- Group 3 - PfSPZ-GA1 Vaccine (Experimental): Group 3 will comprise of 13 volunteers who will receive one immunization of 9.0 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine via DVI.
  Volunteers will be followed closely for monitoring of adverse events and possible breakthrough blood infections by testing for the presence of parasitemia by qPCR. All volunteers will be treated with a curative regimen of atovaquone/proguanil (A/P) should break-through parasites be detected in the peripheral blood, or at the end of the follow-up period (28 days) if they are not qPCR positive. Six months after the inoculation, a final visit will take place to assess adverse events.
  Interventions: Biological: PfSPZ-GA1 Vaccine
- Group 4 - PfSPZ-GA1 Vaccine (Experimental): Group 4 will comprise of 13 volunteers who will receive 3 immunizations of 9.0 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine 8 weeks apart via DVI.
  3 weeks after the last injection, volunteers will undergo mosquito-bite CHMI with five NF54-infected mosquitoes. After CHMI, volunteers will be followed closely for monitoring of adverse events and blood stage infections, and will be seen once daily from day 6 until day 21 after infection and on day 28. All volunteers will be treated with a curative regimen of antimalarials, which may be A/P or artemether/lumefantrine, at the time of detection of blood stage parasitemia by qPCR or 28 days after CHMI. Adverse events will be assessed up to 6 months after the CHMI.
  Interventions: Biological: PfSPZ-GA1 Vaccine; Biological: Mosquito-bite CHMI
- Group 5 - PfSPZ-GA1 Vaccine (Experimental): Group 5 will comprise of 13 volunteers who will receive 3 immunizations of 4.5 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine 8 weeks apart via DVI.
  3 weeks after the last injection, volunteers will undergo mosquito-bite CHMI with five NF54-infected mosquitoes. After CHMI, volunteers will be followed closely for monitoring of adverse events and blood stage infections, and will be seen once daily from day 6 until day 21 after infection and on day 28. All volunteers will be treated with a curative regimen of antimalarials, which may be A/P or artemether/lumefantrine, at the time of detection of blood stage parasitemia by qPCR or 28 days after CHMI. Adverse events will be assessed up to 6 months after the CHMI.
  Interventions: Biological: PfSPZ-GA1 Vaccine; Biological: Mosquito-bite CHMI
- Group 6 - PfSPZ Vaccine (Experimental): Group 6 will comprise of 13 volunteers who will receive 3 immunizations of 4.5 x 10^5 PfSPZ of PfSPZ Vaccine 8 weeks apart via DVI.
  3 weeks after the last injection, volunteers will undergo mosquito-bite CHMI with five NF54-infected mosquitoes. After CHMI, volunteers will be followed closely for monitoring of adverse events and blood stage infections, and will be seen once daily from day 6 until day 21 after infection and on day 28. All volunteers will be treated with a curative regimen of antimalarials, which may be A/P or artemether/lumefantrine, at the time of detection of blood stage parasitemia by qPCR or 28 days after CHMI. Adverse events will be assessed up to 6 months after the CHMI.
  Interventions: Biological: PfSPZ Vaccine; Biological: Mosquito-bite CHMI
- Group 7 - Normal Saline Placebo control (Placebo Comparator): Group 7 will comprise of 9 volunteers who will receive 3 injections of normal saline placebo 8 weeks apart via DVI.
  3 weeks after the last injection, volunteers will undergo mosquito-bite CHMI with five NF54-infected mosquitoes. After CHMI, volunteers will be followed closely for monitoring of adverse events and blood stage infections, and will be seen once daily from day 6 until day 21 after infection and on day 28. All volunteers will be treated with a curative regimen of antimalarials, which may be A/P or artemether/lumefantrine, at the time of detection of blood stage parasitemia by qPCR or 28 days after CHMI. Adverse events will be assessed up to 6 months after the CHMI.
  Interventions: Other: Normal Saline; Biological: Mosquito-bite CHMI

INTERVENTIONS:
Biological: PfSPZ-GA1 Vaccine — Aseptic, purified, cryopreserved, genetically attenuated P. falciparum sporozoites (Pf∆b9∆slarp), strain NF54
  Arms: Group 1 - PfSPZ-GA1 Vaccine; Group 2 - PfSPZ-GA1 Vaccine; Group 3 - PfSPZ-GA1 Vaccine; Group 4 - PfSPZ-GA1 Vaccine; Group 5 - PfSPZ-GA1 Vaccine
Biological: PfSPZ Vaccine — Aseptic, purified, cryopreserved, radiation attenuated P. falciparum sporozoites (PfSPZ Vaccine), strain NF54
  Arms: Group 6 - PfSPZ Vaccine
Other: Normal Saline — 0.9% sodium chloride
  Arms: Group 7 - Normal Saline Placebo control
Biological: Mosquito-bite CHMI — Bites of 5 infected mosquitoes of NF54 strain
  Arms: Group 4 - PfSPZ-GA1 Vaccine; Group 5 - PfSPZ-GA1 Vaccine; Group 6 - PfSPZ Vaccine; Group 7 - Normal Saline Placebo control

SUMMARY:
This is a first-in-human, randomized clinical trial of PfSPZ-GA1 Vaccine (genetically attenuated PfSPZ) in healthy malaria-naïve adult volunteers. This Phase 1 trial is divided into two stages, Stage A and B. Stage A is an open label, single center, dose escalation study in 19 volunteers. Stage B is a multi-center, double blind, randomized, placebo-controlled trial in 48 volunteers. The primary objective of this study is to determine the safety and tolerability of direct venous inoculation (DVI) of PfSPZ-GA1 Vaccine in healthy adults.

DETAILED DESCRIPTION:
Stage A, a Phase 1 dose-escalation study, will take place at Leiden University Medical Centre (LUMC). Stage B, a randomized, double-blind, placebo-controlled trial, will be conducted at LUMC and Radboudumc University Medical Centers (RUMC).

In Stage A, 19 healthy, adult volunteers will be allocated into three groups to receive increasing doses of PfSPZ-GA1 Vaccine by DVI. Group 1 (n=3) will receive one dose of 1.35 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine. If this dose is safe for 28 days after inoculation, then Group 2 (n=3) will receive one dose of 4.5 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine. If this dose is safe for 28 days after inoculation, Group 3 (n=13) will receive one dose of 9.0 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine. Volunteers will be followed closely for monitoring of adverse events and possible breakthrough blood infections by testing for the presence of parasitemia by qPCR. All volunteers will be treated with a curative regimen of atovaquone/proguanil (A/P) should break-through parasites be detected in the peripheral blood, or at the end of the follow-up period (28 days) if they are not qPCR positive. Six months after the inoculation, a final visit will take place to assess adverse events.

If inoculation is deemed safe after 28 days for Group 3 and criteria for proceeding to Stage B are met, the trial will continue to Stage B. In Stage B, 48 healthy, adult volunteers will be randomized into four groups at 2 centers, LUMC and RUMC (24 volunteers at each site). Each group will receive 3 repeat doses, 8 weeks apart, of PfSPZ-GA1 Vaccine (low and high doses), PfSPZ Vaccine (radiation attenuated sporozoites), or normal saline (NS) placebo (as control) via DVI. Group 4 (n=13) will receive 9.0 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine/dose. Group 5 (n=13) will receive 4.5 x 10^5 PfSPZ of PfSPZ-GA1 Vaccine/dose. Groups 6 (n=13) and 7 (n=9) will receive 4.5 x 10^5 PfSPZ Vaccine and NS placebo per dose, respectively. Three weeks after the last inoculation, all immunized volunteers and placebo controls (Group 7) will undergo a CHMI with five NF54-infected mosquitoes (wild-type) to determine degree of protection. After the CHMI, volunteers will be followed closely for monitoring of adverse events and blood stage infections, and will be seen once daily from day 6 until day 21 after infection and on day 28. All volunteers will be treated with a curative regimen of antimalarials, which may be A/P or alternatively artemether/lumefantrine dosed according to Dutch clinical practice, at the time of detection of blood stage parasitemia by qPCR or 28 days after CHMI. Adverse events will be assessed up to 6 months after the CHMI.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 18 and ≤ 35 years and in good health.
* Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
* Subject is able to communicate well with the investigator, is available to attend all study visits.
* Furthermore, the subject will remain within the Netherlands from day -1 till day +28 after each parasite exposure. After CHMI, subjects have to be reachable by phone (24/7) from day -1 until day 35.
* Subject agrees to inform his/her general practitioner (GP) about participation in the study and to sign a request to release by the GP, and medical specialist when necessary, any relevant medical information concerning possible contra-indications for participation in the study.
* Subject agrees to refrain from blood donation to Sanquin or for other purposes throughout the study period and for a defined period thereafter according to Sanquin guidelines (3 years minimum, depending on serology).
* Non-pregnant, non-lactating females of reproductive potential (i.e., have a uterus and are neither surgically sterilized nor post-menopausal) should agree to use adequate contraception and not to breastfeed for the duration of study.
* Subject agrees to refrain from intensive physical exercise (disproportionate to the subjects' usual daily activity or exercise routine) for twenty-one days following each immunization and during the malaria challenge period.
* Subject has signed informed consent.

Exclusion Criteria:

* Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, psychiatric or other disorders, which could compromise the health of the volunteer during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

  1. Body weight < 50 kg or Body Mass Index (BMI) < 18.0 or > 30.0 kg/m^2 at screening
  2. A heightened risk of cardiovascular disease, defined as: i) an estimated ten-year risk of fatal cardiovascular disease of = 5% at screening, as determined by the Systematic Coronary Risk Evaluation (SCORE), ii) history, or evidence at screening, of clinically significant arrhythmia's, prolonged QT-interval or other clinically relevant ECG abnormalities, or iii) a positive family history of cardiac events in first or second degree relatives (according to the system used in medical genetics) < 50 years old
  3. Functional asplenia, sickle cell trait/disease, thalassaemia trait/disease or G6PD deficiency
  4. History of epilepsy in the period of five years prior to study onset, even if no longer on medication
  5. Positive HIV, HBV or HCV screening tests
  6. Chronic use of i) immunosuppressive drugs, ii) antibiotics, or iii) other immune modifying drugs within three months prior to study onset (excluding inhaled and topical corticosteroids and incidental use of oral anti-histamines) or expected use of such during the study period
  7. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past five years
  8. Any history of treatment for severe psychiatric disease by a psychiatrist in the past year
  9. History of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset, positive urine toxicology test for cocaine or amphetamines at screening or prior to infection or positive urine toxicology test for cannabis prior to infection.
* For female subjects: breastfeeding, or positive urine pregnancy test at screening or prior to immunization or prior to CHMI.
* Any history of malaria, positive serology for P. falciparum, or previous participation in any malaria (vaccine) study or CHMI.
* Known hypersensitivity to or contra-indications (including co-medication) for use of atovaquone/ proguanil or artemether/lumefantrine, or history of severe (allergic) reactions to mosquito bites.
* Receipt of any vaccinations in the 3 months prior to the start of the study or plans to receive any other vaccinations during the study period or up to 8 weeks thereafter.
* Participation in any other clinical study in the 30 days prior to the start of the study or during the study period.
* Being an employee or student of the department of Medical Microbiology or Infectious Diseases of the Radboudumc or the LUMC.
* Any other condition or situation that would, in the opinion of the investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol or would compromise the integrity of the data.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Presence of blood stage parasites after inoculation with PfSPZ-GA1 Vaccine in Stage A | From time of inoculation to till 28 days later
  Presence of blood stage parasites after inoculation with PfSPZ-GA1 vaccine, as assessed by qPCR
Frequency and magnitude of adverse events in study groups in Stage A and B | From time of inoculation to end of study, assessed up to 17 months
  Frequency and magnitude of adverse events in study groups

SECONDARY OUTCOMES:
Presence of parasitemia after CHMI in Stage B | From time of inoculation to till 28 days later
  Presence of parasitemia after CHMI with the wild-type NF54 strain, as detected by qPCR

CONTACTS AND LOCATIONS:
Overall Officials: Robert W. Sauerwein, MD, Principal Investigator — Radboud University Medical Center, Geert Grooteplein 28, 6525 GA Nijmegen, The Netherlands; Leo G Visser, MD, Principal Investigator — Leiden University Medical Center, Albinusdreef 2, 2333 ZA Leiden, The Netherlands
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Albinusdreef 2, Leiden
  - Radboud University Medical Center, Geert Grooteplein 28, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Schaijk BC, Ploemen IH, Annoura T, Vos MW, Foquet L, van Gemert GJ, Chevalley-Maurel S, van de Vegte-Bolmer M, Sajid M, Franetich JF, Lorthiois A, Leroux-Roels G, Meuleman P, Hermsen CC, Mazier D, Hoffman SL, Janse CJ, Khan SM, Sauerwein RW. A genetically attenuated malaria vaccine candidate based on P. falciparum b9/slarp gene-deficient sporozoites. Elife. 2014 Nov 19;3:e03582. doi: 10.7554/eLife.03582. PMID 25407681